CLINICAL TRIAL: NCT06089395
Title: A Randomized and Double-blind Clinical Trial of Jiajian Guishen Granules on the Modulation of Ovarian Function in Patients With Poor Ovarian Response
Brief Title: The Effect of Jiajian Guishen Granules on the Modulation of Ovarian Function in Patients With Poor Ovarian Response(POR)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shi Yun (Other)
Collaborators: Capital Medical University (Other)
Responsible Party: Sponsor-Investigator, Shi Yun, Chief of Gynecology, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JJGS on POR
Record Dates: First submitted 2023-10-04; First posted 2023-10-18 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Poor Ovarian Response
Keywords: Poor Ovarian Response; Ovarian function; Jiajian Guishen granules
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Intervention Model Description: A Stratified Block Group Randomized Controlled Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jiajian Guishen granules group (Experimental): Jiajian Guishen granules + coenzyme Q10 simulant
  Interventions: Drug: Jiajian Guishen granules
- coenzyme Q10 group (Active Comparator): Jiajian Guishen granules simulant+ coenzyme Q10
  Interventions: Drug: coenzyme Q10

INTERVENTIONS:
Drug: Jiajian Guishen granules — This study was a stratified district group randomized, double-blind, double simulation, positive control clinical trial with JJGS granules + coenzyme Q10 simulant in the test group and JJGS granules simulant + coenzyme Q10 in the control group
  Other Names: JJGS
  Arms: Jiajian Guishen granules group
Drug: coenzyme Q10 — This study was a stratified district group randomized, double-blind, double simulation, positive control clinical trial with JJGS granules + coenzyme Q10 simulant in the test group and JJGS granules simulant + coenzyme Q10 in the control group
  Other Names: CoQ10
  Arms: coenzyme Q10 group

SUMMARY:
Relying on the Department of Gynecology of Dongzhimen Hospital of Beijing University of Traditional Chinese Medicine and chaoyang hospital of Capital medical university, this randomized controlled clinical study was carried out to investigate the application of kidney tonifying herbs to patients with poor ovarian response（POR）.

A total of 76 patients with POR were collected and stratified district groups were randomly divided into a test group and a control group, with 38 patients included in each group. The experimental group was intervented with JJGS granules + coenzyme Q10 simulant, and the control group was intervened with coenzyme Q10 + JJGS granules simulant. AMH, serum basal sex hormone, AFC, TCM syndrome score, modified Kupperman scale and pregnancy status were observed before and after treatment to investigate the effects of Jiajian Guishen granules on the ovarian function of POR patients.

DETAILED DESCRIPTION:
This study was a multicenter, stratified block randomized, double-blind, double simulation, positive controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Woman who meet the diagnostic criteria for poor ovarian response;
2. Woman who meet the TCM diagnostic criteria for kidney deficiency;
3. Woman whose serum basal FSH(two consecutive menstrual cycles)between 10-25mIU/mL
4. Woman whose AMH <1.1ng/ml;
5. Woman aged ranged from 20-45 years old
6. Woman whose body mass index (BMI)<35 kg/m2
7. Womanwho voluntarily signed the informed consent form.

Exclusion Criteria:

1. Woman who have combination of serious diseases such as cardiovascular, cerebrovascular, hepatic, renal and hematopoietic systems, and malignant tumors;
2. Woman who have other endocrine diseases, such as polycystic ovary syndrome and hyperprolactinemia;
3. Woman who are unable to cooperate with the treatment and follow-up, such as combined neurological and psychiatric disorders, or those who are unwilling to cooperate.
4. Woman who have used the same efficacy of herbs or other therapies in the last 1 month;
5. Woman who are allergic to the drugs used in this study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Anti-Miller's Tube Hormone（AMH） | before treatment and the first menstrual period 2-4 days after treatment
  The unit is ng/mL.Elbow vein blood was collected on an empty stomach, and after separating the serum, anti-mullerian hormone (AMH) was measured by radioimmunoassay

SECONDARY OUTCOMES:
Follicle-stimulating hormone（FSH） | before treatment and the first menstrual period 2-4 days after treatment
  The unit is mIU/mL.Elbow vein blood was collected on an empty stomach, and after separating the serum, FSH were measured by radioimmunoassay.
Luteinizing hormone（LH） | before treatment and the first menstrual period 2-4 days after treatment
  The unit is mIU/mL.Elbow vein blood was collected on an empty stomach, and after separating the serum, LH were measured by radioimmunoassay.
Estrogen (E2) | before treatment and the first menstrual period 2-4 days after treatment
  The unit is pg/mL.Elbow vein blood was collected on an empty stomach, and after separating the serum, E2 were measured by radioimmunoassay.
Progesterone (P) | before treatment and the first menstrual period 2-4 days after treatment
  The unit is ng/mL.Elbow vein blood was collected on an empty stomach, and after separating the serum, P were measured by radioimmunoassay.
Testosterone（T） | before treatment and the first menstrual period 2-4 days after treatment
  The unit is ng/mL.Elbow vein blood was collected on an empty stomach, and after separating the serum, T were measured by radioimmunoassay.
antral follicle count（AFC） | before treatment and early follicular phase in the first post-treatment menstrual cycle day 1
  Color Doppler ultrasound was performed in the early follicular phase in the usual way to observe the number of follicles in the underlying sinuses.
Traditional Chinese Medicine Score | baseline and immediately after treatment
  The main symptoms include menstrual cycle, menstrual flow reduction. Scoring criteria: ① normal menstrual cycle 0 points, 1-2 weeks ahead or behind the wrong 4 points, 2-3 weeks 8 points, more than 3 weeks 12 points; ② menstrual flow than the previous menstrual flow no change 0 points, menstrual flow reduction ≤ ⅓ 4 points, ⅓ < menstrual flow reduction ≤ ½ 8 points, menstrual flow reduction > ½ 12 points. Secondary symptoms included lumbar and knee pain, dizziness and tinnitus, loss of libido, increased urination, hot flashes and night sweats, and lower back and lower limb pain. According to the degree of aggravation of symptoms, the total score was assigned as 0,2,4,8. The sum of the scores of the main symptoms and secondary symptoms, the higher the score, the more serious the TCM symptoms.
Modified Kupperman rating scale | baseline and immediately after treatment
  Referring to the domestic modified Kupperman Symptom Scoring Criteria in Chinese Obstetrics and Gynecology, edited by Cao Zeyi, to observe and rate perimenopausal symptoms before and after treatment and to quantify the degree of decline in ovarian function.Entries include hot flashes and sweating, sensory abnormalities, insomnia, anxiety and depression, dizziness, fatigue, muscle and joint pain, headache, palpitations, ankylosis of the skin, sexual discomfort, and urinary irritation, with different coefficients for each entry, and according to the aggravating degree of the symptom, they are divided into 0, 1, 2, and 3 points, and the coefficients corresponding to the scoring of the degree of each item are multiplied by a fixed score of the symptom to add up to the total score, and the higher the total score suggests that the symptoms of the perimenopausal period are more serious.
Clinical pregnancy rate | up to 6 months
  Defined as the number of women with identified clinical pregnancies divided by the number of patients randomized to a specific group. Clinical pregnancy is confirmed when 1 or more ges-tational sacs are detected on transvaginal ultrasound assessment.
Early miscarriage rate | up to 6 months
  Defined as the per-centage of participants with loss of a diagnosed clinical pregnancy before 12 weeks gestation to the total patients randomized

CONTACTS AND LOCATIONS:
Overall Officials: Shi Y Shi Yun, phD, Study Director — Dongzhimen Hospital of Beijing University of Chinese Medicine; Wang CM Wang Chunmei, phD, Principal Investigator — Dongzhimen Hospital of Beijing University of Chinese Medicine; Shi X Shi Xiao, phD, Principal Investigator — Capital Medical University; Yang QH Yang Qiaohui, pdD, Principal Investigator — Dongzhimen Hospital of Beijing University of Chinese Medicine; Yan QY Yan Qingya, phD, Principal Investigator — Dongzhimen Hospital of Beijing University of Chinese Medicine; Shao JY Shao Jingyi, Master, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine; Xu K Xu Ke, Master, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine; Li XY Li Xiyu, Bachelor, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine; Liu QY Liu Qinyang, Bachelor, Study Chair — Dongzhimen Hospital of Beijing University of Chinese Medicine
Locations (2):
- China (2):
  - Dongzhimen Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Chaoyang Hospital Affiliated to Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
We will share the protocol and progress of the clinical trial, and will share the clinical study report when we have completed patient collection and treatment.
Supporting Information: Study Protocol, CSR
Time Frame: IPD is available from Aug 2025 for 5 years
Access Criteria: All investigators can check through the public management platform of clinical trials, or contact the investigators of this trial to obtain IPDs including clinical trial protocols and clinical trial reports.
URL: https://www.dzmyy.com.cn/